CLINICAL TRIAL: NCT00299910
Title: Inflammatory Response to Anti Inflammatory Therapy in Children With Sleep Disordered Breathing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sor388505ctil
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — montelukast

INTERVENTIONS:
Drug: Montelukast

SUMMARY:
This study will assess in a double blind placebo controlled fashion the effects of a 12 week course of oral montelukast/placebo on polysomnographic and radiological findings and will characterize the systemic (serum,urine) and local (upper airway collected biological samples) inflammatory response in children (2-10 years of age) with sleep disordered breathing, fittingthe inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:2-10 years old

1<AHI<8 measured in an overnight PSG

-

Exclusion Criteria:

Asthma Previous use or allergy to montelukast Use of antibiotics in the previous 3 weeks Use of corticosteroids in the previous 3 months Craniofacial dysmorphism Genetic or metabolic defined illnesses Adenotonsillectomy or adenoidectomy in the past

-

Ages: 2 Years to 10 Years | Sex: All
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Pediatric Sleep Center, Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Goldbart AD, Goldman JL, Veling MC, Gozal D. Leukotriene modifier therapy for mild sleep-disordered breathing in children. Am J Respir Crit Care Med. 2005 Aug 1;172(3):364-70. doi: 10.1164/rccm.200408-1064OC. Epub 2005 May 5. PMID 15879419